



# PROspective multiethnic validation of the BEhçet's syndrome Overall Damage Index (BODI): the PROBE study



# **INDEX**

| Administrative Information | PAG. 3 |
|-----------------------------|---------|
| Roles and Responsibilities | PAG.4 |
| Background | PAG.6 |
| OBJECTIVES | PAG. 6 |
| METHODS | PAG.7 |
| STUDY TIMELINE | PAG. 13 |
| Publication Rules | PAG. 14 |
| ETHIC AND REGULATORY ISSUES | PAG. 14 |
| References | PAG. 17 |



## **ADMINISTRATIVE INFORMATION**

## TITLE:

PROspective multiethnic validation of the BEhçet's syndrome Overall Damage Index (BODI): the PROBE study

| Data Category | Information |
|---|---|
| Primary registry and study identifying number | In progress |
| Date of registration in primary registry | In progress |
| Source(s) of monetary or material support | No funding |
| Primary sponsor | NA |
| Secondary sponsor(s) | NA |
| Contact for public queries | matteopiga@unica.it |
| Contact for scientific queries | bodiproject@gmail.com |
| Public title | PROBE study |
| Scientific title | PROspective multiethnic validation of the BEhçet's syndrome Overall Damage Index (BODI): the PROBE study |
| Countries of recruitment | Worldwide |
| Health condition studied | Behçet' syndrome |
| Study design | Observational study |

PROTOCOL VERSION: 1.0

| Issue Date: | 25 March 2021 |
|----------------------------|-------------------------------------------|
| Protocol amendment number: | 1 |
| Author(s): | Matteo Piga, Alberto Floris, Gülen Hatemi |

## **CONFIDENTIALITY STATEMENT**

The information contained in this document is the property of the University of Pisa and therefore is provided to you in confidence for review by you, your staff, an applicable Ethics Committee/Institutional Review, and regulatory authorities. It is understood that the information will not be disclosed to others without prior written approval except to the extent necessary to obtain informed consent from those persons to whom the medication may be administered.



LIST OF THE INVOLVED RESEARCH CENTRES AND ROLES AND RESPONSIBILITIES OF INVESTIGATORS

| | Research Centres | Investigators' name and role |
|---|---|---|
| 1. | Rheumatology Unit, University and AOU of Cagliari,<br>Monserrato – Italy (Proposing and coordinating Centre) | Matteo Piga (Italy)<br>Principal Investigator |
| | | Alberto Cauli (Italy)<br>Executive committee |
| | | Alberto Floris (Italy)<br>Executive committee |
| 2. | Department of rheumatology National Reference<br>Centre for Rare Auto-Immunes Diseases, Hôpital de<br>Hautepierre, Strasbourg Cedex, France | Laurent Arnaud (France) Executive committee |
| 3. | Université des Sciences et de la Technologie Houari<br>Boumediene: Algiers | Houda Belguendouz (Algeria)<br>Investigator |
| 4. | Department of Rheumatology, Clinical Immunology and Allergy, University of Crete School of Medicine - Greece | George Bertsias (Greece)<br>Investigator |
| 5. | Department of Rheumatology, Mayo Clinic, Jacksonville, Florida - USA | Ronald Butendieck (USA)<br>Investigator |
| 6. | Rheumatology Unit, University of Siena. Policlinico Le<br>Scotte, Siena - Italy | Luca Cantarini (Italy)<br>Investigator |
| 7. | Department of Autoimmune Diseases, Hospital Clinic, IDIBAPS, University of Barcelona - Spain | Ricard Cervera (Spain)<br>Investigator |
| | | Gerard Espinosa (Spain)<br>Investigator |
| 8. | Clinical Immunology Unit, Centro Hospitalar do Porto and UMIB, ICBAS, Universidade do Porto, Portugal. | Joao Correja (Portugal)<br>Investigator |
| | | Carlos Vasconcelos (Portugal)<br>Investigator |
| 9. | Ophthalmology Unit, Department of Medical Sciences,<br>Surgery and Neurosciences, University of Siena , Italy | Claudia Maria Fabiani (Italy)<br>Investigator |
| 10 | Department of Medical Sciences, Section of Rheumatology, AOU S. Anna, University of Ferrara - Italy | Marcello Govoni (Italy)<br>Investigator |
| 11 | Department of Internal Medicine, Division of Rheumatology, Istanbul University - Cerrahpasa | Gülen Hatemi (Turkey)<br>Investigator |



| Research Centres | Investigators' name and role |
|---|---|
| 12. University of Tunis El Manar, Faculty of Medicine of Tunis, LR99ES11 Tunis, Tunisia; Rabta Hospital, Service of Internal Medicine, Jebbari 1007, Tunis, Tunisia. | Habib Mohamed Houman<br>(Tunisia)<br>Investigator |
| 13. Connective Tissue Diseases Research Center, Tabriz University of Medical Sciences, Tabriz, Iran. | Alireza Khabbazi (Iran)<br>Investigator |
| 14. Department of Dermatology, Severance Hospital,<br>Cutaneous Biology Research Institute, Yonsei University<br>College of Medicine, Seoul, Korea | Do Young Kim (South Korea) Investigator |
| 15. Department of Emergency and Organ Transplantation,<br>Rheumatology Unit, University of Bari - Italy | Florenzo Iannone (Italy)<br>Investigator |
| 16. Department of Medicine, Nazarbayev University School of Medicine (NUSOM), Nur-Sultan, Kazakhstan. | Dimitri Poddighe (Kazakhstan)<br>Investigator |
| 17. Internal Medicine Department, Rheumatology and Clinical Immunology Unit, Faculty of Medicine, Cairo University, Cairo, Egypt. | Gaafar Ragab (Egypt)<br>Investigator |
| 18. Sorbonne Universités AP-HP, Groupe Hospitalier Pitié-<br>Salpêtrière, Département de Médecine Interne et<br>Immunologie Clinique, Paris, France. | David Saadoun (France)<br>Investigator |
| 19. Division of Rheumatology, Universidade Federal de São Paulo, São Paulo, Brazil. | Alexandre WS de Souza (Brazil)<br>Investigator |
| 20. Department of Immunology, School of Medicine, Tehran University of Medical Sciences, Tehran, Iran. | Farhad Shahram (Iran)<br>Investigator |
| 21. Department of Rheumatology, Peking Union Medical College Hospital, Beijing, China | Wenjie Zheng (China)<br>Investigator |
| 22. Internal Medicine Department, Ibn Sina University Hospital, Rabat, Morocco. | Tazi Mezalek Zoubida (Moroc)<br>Investigator |



#### **BACKGROUND**

Behçet's syndrome (BS) is a multisystem inflammatory disease of unknown etiology, characterized by strong genetic background, distinctive geographic distribution, and wide variability in clinical presentation [1]. Disease activity related to BS as well as chronic exposure to medications may lead to the development and accrual of irreversible organ damage resulting in impairment of quality of life, disability, and increased mortality [2]. For these reasons, organ damage was included in the OMERACT outcome core set for BS [3].

The Behçet's syndrome Overall Damage Index (BODI) is a recently developed tool to identify and measure organ damage in BS [2]. The BODI is grounded in a solid evidence-based and consensus-based methodology, and its preliminary validation on a multicenter cohort of Southern European patients showed highly promising performance in terms of comprehensiveness, specificity, reliability, sensitivity to change, and feasibility [2].

Nevertheless, a prospective validation with a wider and ethnically heterogeneous cohort of BS patients is needed to generally evaluate the impact of those BODI items seldom recorded or absent in the preliminary validation cohort and to weigh the damage items depending on their relevance for predicting major outcomes.

#### **OBJECTIVES**

## **General objectives**

The general objectives of the PROBE study are to further test the comprehensiveness of the BODI (content validity) in a wide and ethnically heterogeneous cohort of BS patients, and investigate how damage assessed by the BODI correlates with other major long-term disease outcomes (criterion validity), with the ultimate goal of drafting a weighing system for each BODI item.

## **Specific Objectives**

- 1. To test the comprehensiveness of the instrument in a wide and ethnically heterogeneous cohort of BS patients, evaluating the prevalence of those BODI items seldom recorded or absent in the preliminary validation cohort
- 2. To describe possible differences in the entity and type of damage accrual in BS patients from different geographical areas.
- 3. To identify the factors independently associated with damage development and accrual.



- 4. To investigate the association between the results of the baseline BODI measurement (BODI ≥1, BODI score, and BODI ranking) and the 5-years mortality rate.
- 5. To investigate the association between the results of the baseline BODI measurement (BODI ≥1, BODI score, and BODI ranking)and the 5-years hospitalization rate.
- 6. To weigh each item of damage depending on their relevance in predicting mortality.

#### **METHODS**

## Study design

PROBE is an observational multicenter cohort study, consisting of a cross-sectional and a 5-years prospective phase, designed to target the major study objectives, such as testing the content and criterion validity of the BODI and drafting a weighing system for each BODI items.

During the study, patients will undergo a routine clinical assessment, as scheduled in their follow-up program. No further clinical, laboratory or instrumental investigations are required in addition to those provided according to good clinical practice. Treatment prescription will be evaluated by each investigator independently from the study and according to the international and local guidelines and the good clinical practice.

#### **Patients**

The study population will consist of <u>consecutive</u> BS patients diagnosed according to the ICBD or ISG classification criteria [4,5] recruited in Centers with expertise for BS.

## **Inclusion criteria**:

Diagnosis of BS according to ICBD or ISG criteria;

## **Exclusion criteria:**

 subjects unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow interval visits.

Any effort should be addressed by investigators to minimize the rate of lost to follow-up and guarantee the completeness of the database.



#### **Data collection**

Data will be collected at the time of recruitment (baseline, T0) and then annually (± 1 month) for 5 years. Overall, 6 visits are planned to be recorded (T0, T1, T2, T3, T4, T5). Details on the data required at each visit are reported in table 1.

A query management system (QMS) will manually track data queries so they can be adequately individualized and resolved. QMS substantially minimizes and even eliminates the risk of invalid data being unnoticed. Collected data will be checked annually and data queries (e.g., data issue) will be forwarded to Investigators. Data queries will only be resolved in the following ways:

- by correcting the error, in other words entering a new value that is valid;
- by marking the data in conflict as correct.

Table 1. Data collection at each scheduled visit

| Table 1. Data collection at each schedule | TO | T1 | T2 | Т3 | <b>T4</b> | T5 |
|---|---|---|---|---|---|---|
| Months | Baseline | 12 (±1) | 24 (±1) | 36 (±1) | 48 (±1) | 60 (±1) |
| Demographics | Р | | | | | |
| Comorbidities | Р | | | | | |
| Cumulative disease manifestations | Р | | | | | |
| Active manifestations between visits | | Р | Р | Р | Р | Р |
| BD current activity form (BDCAF) | Р | Р | Р | Р | Р | Р |
| BODI score | Р | Р | Р | Р | Р | Р |
| Physician global assessment (PGA) | Р | Р | Р | Р | Р | Р |
| Patient's global assessment (PtGA) | Р | Р | Р | Р | Р | Р |
| Patient's damage assessment (PtDA) | Р | Р | Р | Р | Р | Р |
| Ongoing treatment | Р | Р | Р | Р | Р | Р |
| N of relapses (between visits) | Last 5 yrs | Р | Р | Р | Р | Р |
| N of hospitalizations (between visits) | Last 5 yrs | Р | Р | Р | Р | Р |
| Death | | Р | Р | Р | Р | Р |



## **Variables**

Details on the variables that are requested to be recorded are reported below:

## • Demographics:

- o Gender (male/female)
- o Date of birth
- o Date of onset:
  - a) first disease manifestation including oral aphtosis;
  - b) first disease manifestation excluding oral aphtosis
- o Date of diagnosis
- Date of enrolment
- Smoking:
  - never smoker,
  - current smoker,
  - past smoker
- o Country of origin
- Country of residence
- Ethnicity:
  - Caucasian;
  - Asian;
  - Hispanic;
  - Afro-American;
  - Arab;
  - Other (please specify)
- o Education level:
  - Illiterate
  - Primary school
  - Secondary School
  - College/University

## Comorbidities:

- Fibromyalgia
- Blood hypertension



- Dyslipidemia
- Obesity (BMI>30)
- Chronic Kidney disease
- Diabetes (diagnosed before onset of BS)
- Other (please specify)
- Cumulative clinical manifestations: any disease manifestation occurred from the disease onset to the enrolment visit (even no longer present at the enrolment visit). The following disease manifestations have to be recorded:
  - Oral aphtosis (yes/no)
  - Genital aphtosis (yes/no)
  - Skin lesions (yes/no, if yes specify which type)
  - Ocular (yes/no, if yes specify which type)
  - Vascular (yes/no, if yes specify which type)
  - Neurologic (yes/no, if yes specify which type)
  - Musculoskeletal (yes/no, if yes specify which type)
  - Gastrointestinal yes/no, (if yes specify which type)
  - Pathergy test (yes/no)
  - Others yes/no, (if yes specify which type)
- Active clinical manifestations between visits: manifestations that are present at the time of the visit or have occurred since last visit. The following disease manifestations have to be recorded:
  - Oral aphtosis (yes/no)
  - Genital aphtosis (yes/no)
  - Skin lesions (yes/no, if yes specify which type)
  - Ocular (yes/no, if yes specify which type)
  - Vascular (yes/no, if yes specify which type)
  - Neurologic (yes/no, if yes specify which type)
  - Musculoskeletal (yes/no, if yes specify which type)
  - Gastrointestinal yes/no, (if yes specify which type)
  - Pathergy test (yes/no)
  - Others yes/no, (if yes specify which type)



- Behçet's disease current activity form (BDCAF) score: BDCAF is a disease activity assessment tool for BS. It depends on an accurate evaluation of clinical features present during the month before the date of assessment. The presence/absence of 9 somatic symptoms from a list may be recorded, together with eye involvement, nervous system involvement, major vessel involvement, as well as the clinician's overall perception of disease activity. The transformed index score on an interval scale will be used for analysis in the present study. [6]
- Behçet's syndrome overall damage index (BODI). It is a tool recently developed to identify and measure organ damage in BS. BODI consists of 4 overarching principles and 34 items with 12 subitems, categorized into 9 organ/system domains: mucocutaneous, musculoskeletal, ocular, vascular, cardiovascular, neuropsychiatric, gastrointestinal, reproductive system, and miscellaneous. Each item and subitem scores 1 point. The total score ranges from 0 to 46 [2]. In order to score the BODI, each investigator will be provided with a user manual and a video tutorial (https://vimeo.com/264992929).
- Physician's global assessment of disease activity (PGA). It will be assessed through a single question ("How active is the patient's BS?") on an anchored 10-cm visual analogic scale (0.5-cm graded), where 0 corresponded to "no disease activity" and 10 to "the highest disease activity." [7]
- Patient's global assessment of disease activity (PtGA). It will be assessed through a single question ("How active was your BS during the last week?") on an anchored 10-cm visual analogic (0.5-cm graded), where 0 corresponded to "no disease activity" and 10 to "the highest disease activity." [7]
- Patient's damage assessment (PtDA). It will be assessed through a single question ("How much irreversible (non-healing) damage have you developed since the diagnosis of BS?") on an anchored 10-cm visual analogic (0.5-cm graded), where 0 corresponded to "no damage" and 10 to "the highest amount of damage".
- Ongoing treatment: medications that are ongoing at the time of each visit will be classified
   as:
  - Colchicine (yes/no)



- Glucocorticoids (yes/no, if yes specify the current dosage in mg/day of prednisone ore equivalents)
- Conventional immunosuppressant (yes/no, if yes which agent; i.e., azathioprine, cyclosporine, cyclophosphamide, thalidomide, methotrexate, sulphasalazine; others)
- Apremilast (yes/no)
- Biologic immunosuppressant (yes/no, if yes which agent; i.e. anti-TNFalpha agents)
- Other (yes/no, if yes specify)
- Number of relapses. Relapse is defined as the onset of a new BS manifestation or recurrence/worsening of a pre-existing clinical manifestation resulting in significant treatment modifications. Significant treatment modifications will be defined as the starting or increasing dosage of corticosteroids, colchicine, apremilast, conventional or biologic immunosuppressant. For each relapse, the clinical manifestation inducing the treatment modification will be recorded.
- **Number of hospitalizations.** Hospitalization will be defined as any admission to the hospital (duration at least one day including emergency room) for any reason both related to BS (i.e. treatment, management of complications, diagnosis of new manifestations, etc.) and unrelated to BS (i.e. surgery, cardiovascular disease, malignancy, etc.). Primary reasons and numbers of days of hospitalization will be recorded.
- Death (yes/no, date of death, cause of death). In this regard, it is of extreme importance to
  make every possible effort to ensure that patients resulting lost to follow-up have not
  deceased.

## **Statistical analysis**

Descriptive statistics will be performed to report on the prevalence and amount of damage, as assessed by the BODI. In the whole study cohort and different geographical sub-groups, the damage will be described as:

- prevalence of any damage (BODI ≥1);
- prevalence of any damage in the different BODI domains;
- mean (SD) or median (IQR) BODI score;

**PROBE** 

ranking of the BODI score will be developed, using a multistate model, depending on the

distribution of damage in the whole population.

Univariate and multivariate regression models will be implemented to investigate the significant

difference between ethnic/geographic groups in terms of prevalence and amount of damage

accrual. Similarly, univariate and multivariate regression models will be implemented to investigate

independent factors associated with the development or accrual of damage, as assessed by the

BODI.

Multivariate Cox proportional hazards regression models will be created to assess the effect of

damage (BODI score, BODI ≥1, BODI ranking) on subsequent risk of death with adjustment for

covariates, including gender, age, disease duration at enrollment, history of major organ

involvement, disease activity at enrolment, comorbidities (onset before BS diagnosis). Results will

be presented as hazard ratios with their corresponding 95% confidence intervals. Statistical

significance will be defined as a P-value <0.05. Finally, adjusted survival estimates obtained from

these Cox regression models were plotted as survival curves.

Sample size

According to the results of previous studies, 95% overall 5-year survival is expected [8]. Assuming

99% and 95% of survival rate in BS patients with and without BODI damage, respectively, and

assuming 50% prevalence of damage (BODI ≥1) in the study cohort, we estimated a required sample

size of at least 801 BS patients (alpha type I error = 0.05; beta type II error 0.20) to identify damage

as a predictor of mortality. Under the assumption of 25%maximum attrition (5% every year), the

sample size will be increased to 1040 patients.

**STUDY TIMELINE** 

March 2021 – June 2021: Investigators involvement and Ethic Approval (if locally required)

April 2021 – December 2021: Enrollment window

January 2022 – December 2026: Prospective follow-up window

**Publication plan:** 

**End of 2022 :** Publication of Cross-sectional results (content validity)

End of 2025: Publication of mid-term results (factors associated to damage accrual)



End of 2028: publication of prospective results (construct validity)

#### **PUBLICATION RULES**

Baseline data will be published in a peer-reviewed scientific journal within 1 year from the end of recruitment. The full results of the prospective validation will be published in a peer-reviewed scientific journal following the completion of the 5-year study. Partial or preliminary results can be published beforehand.

The main publication is the responsibility of the Principal Investigator. Authorship in the main publications, as well as in ancillary papers, will be offered to all Investigators who achieve the minimum target of 30 patients with complete clinical data after 5 years of follow-up. All the other Investigators not reaching these criteria will be included in the collaborator's list according to the table below. Any exception could be evaluated, depending on the number of enrolled patients with complete data, by taking into account the national epidemiological distribution of BS. Investigators will be listed in authorship according to the number (from highest to lowest) of enrolled patients.

| Number of patients | Investigator | Local co-investigator |
|--------------------|--------------|-----------------------|
| >100 | Author | Author |
| 30-100 | Author | Collaborator |
| <30 | Collaborator | Collaborator |

A list of ancillary publications will be discussed; the study proponent will be granted to access the entire data-set and will lead the ancillary publication. Authorship of ancillary papers will be the same as the main publications.

## **ETHIC AND REGULATORY ISSUES**

## **Ethical Committee Approval**

Ethical Committee Approval will be obtained by the Proposing and Coordinating Centre (Rheumatology Unit, AOU of Cagliari, Italy) and in the other Research Centres in accordance with the policy of the Institutions and local legislation for this kind of study.

Any future change to the protocol or informed consent needed over the study must be approved by Ethical Committee.



#### **Data Collection**

Demographic, clinical and therapeutic data will be collected during the enrolment visit and annually for 5 years during the routinary follow-up visits for each patient, by reviewing medical records and clinical files. No further clinical, laboratory or instrumental investigations will be performed in addition to those provide by the good clinical practice. No experimental drugs will be administrated. Any possible drug administration will be evaluated independently to the study and according to the good clinical practice and the observational nature of the study.

## Data entry and security

The collected data from each Research Centre will be anonymously recorded in an electronic spreadsheet. Anonymous data form each Research Centre will be subsequently entered into a single password-protected database managed and guarded by the Coordinating Research Centre (Rheumatology Unit, AOU of Cagliari, Italy). To guarantee anonymity, an alphanumeric code will be attributed to each patient by the recruiting physician. The correspondence between the alphanumeric code and the patient's identity will be reported in a sperate document, accessible only to the recruiting physician. Access to patient final database will be restricted to the Chief Investigator and Collaborators above.

#### Informed consent

The recruiting physician must inform patients on every aspect of the study, including his right to withdraw at any time. The decision of participating to the study must be voluntary.

In accordance with the policy of the Institutions and local legislation of each Research Centre for this kind of study, a signed informed consent will be obtained at the enrolment and a copy of will be provided to the recruited patient also. The informed consent will be signed by the recruiting physician also.

## Study withdrawal

Every recruited patient can withdrawal from the study at any time for any reason. If his data yet entered in the database and not published, they will be removed.



## Data publication and privacy

Following completion of the study, the full results will be published in a peer-reviewed scientific journal. The data anonymity will be guaranteed in accordance with the personal data protect laws.

#### Insurance cover

For the purely observational nature of the study, no further insurance coverage should be requested in addition to that provided for the standard clinical practice by each Research Centre.

## **Funding**

No specific funding is provided for the study

#### **REFERENCES**

- 1. Yazici H, Seyahi E, Hatemi G, Yazici Y. Behçet syndrome: a contemporary view. Nat Rev Rheumatol. 2018;14:107–19.
- 2. Piga M, Floris A, Espinosa G, Pinto LS, Kougkas N, Monaco AL, et al. Development and preliminary validation of the Behçet's syndrome Overall Damage Index (BODI). RMD Open. BMJ Specialist Journals; 2020;6:e001192.
- 3. Hatemi G, Meara A, Ozguler Y, Direskeneli H, Mahr A, Shea B, et al. The OMERACT Core Set of Domains for Outcome Measures in Behçet Syndrome. Arthritis Care Res. 2020;
- 4. Davatchi F, Assaad-Khalil S, Calamia KT, Crook JE, Sadeghi-Abdollahi B, Schirmer M, et al. The International Criteria for Behçet's Disease (ICBD): a collaborative study of 27 countries on the sensitivity and specificity of the new criteria. J Eur Acad Dermatol Venereol. 2014;28:338–47.
- 5. Criteria for diagnosis of Behçet's disease. International Study Group for Behçet's Disease. Lancet Lond Engl. 1990;335:1078–80.
- 6. Bhakta BB, Brennan P, James TE, Chamberlain MA, Noble BA, Silman AJ. Behçet's disease: evaluation of a new instrument to measure clinical activity. Rheumatology. 1999;38:728–33.
- 7. Floris A, Espinosa G, Serpa Pinto L, Kougkas N, Lo Monaco A, Lopalco G, et al. Discordance between patient and physician global assessment of disease activity in Behçet's syndrome: a multicenter study cohort. Arthritis Res Ther. 2020;22:278.
- 8. Saadoun D, Wechsler B, Desseaux K, et al. Mortality in Behçet's disease. Arthritis Rheum 2010;62:2806–12.